CLINICAL TRIAL: NCT03149315
Title: Inhibition of Anaphylaxis by Ibrutinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Principal Investigator, Melanie c Dispenza, MD, PhD, Assistant Professor of Medicine, Northwestern University Feinberg School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-357
Record Dates: First submitted 2017-05-05; First posted 2017-05-11 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Food Allergy; Anaphylaxis Food
MeSH Terms: conditions — Food Hypersensitivity | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Administration (Experimental): Allergic subjects will be given ibrutinib 420mg daily for 2-7 doses to determine the shortest amount of time and fewest ibrutinib doses required to suppress food skin prick testing and basophil activation test reactivity.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib 420mg, PO once daily for 2-7 days
  Other Names: Ibruvica

SUMMARY:
This is a phase II open label study on the use of Ibrutinib on the inhibition of food-induced anaphylaxis in adults with food allergy. Ibrutinib (brand name Imbruvica) is currently FDA approved for the treatment of mantle cell lymphoma (MCL), chronic lymphocytic leukemia (CLL), and Waldenstrom's macroglobulineia (WM). We propose to administer this approved drug to adults with food allergy to inhibit food allergy responses.

DETAILED DESCRIPTION:
This is open-label study designed to determine the fewest doses and shortest length of time, from two days to up to 7 days, needed for ibrutinib to fully inhibit tests for food allergy, and to determine the length of persistence of efficacy after the drug is stopped.

ELIGIBILITY:
Inclusion Criteria:

* History of food allergy to peanut (or tree nut).
* Male or female age ≥ 18 years.
* Positive skin prick testing and basophil activation test to the trigger food, either peanut or tree nut.
* Adequate organ and marrow function as defined below:
* leukocytes ≥ 3,000/mcL
* absolute neutrophil count ≥ 1,500/mcL
* platelets ≥ 100,000/mcl
* total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SPGT) within normal institutional limits
* Creatinine within normal institutional limits
* Women of child bearing potential must agree to two forms of highly effective contraception (hormonal, device, or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform the Principal Investigator and her treating physician immediately.
* A female of child bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent.
* Ability to clearly understand and speak English at an 8th grade reading level. For safety reasons, subjects must speak English due to the anticipated need for clear and timely communication with investigators and the study team in emergency situations, since the investigators and study team are English speaking.

Exclusion Criteria:

* Subjects who have been on immunomodulatory therapies or oral corticosteroids within 1 month prior to study participation will be excluded, and those taking antihistamines must stop these drugs for one week prior to enrollment and must refrain from taking antihistamines during the duration of the study so as not to interfere with SPT responses.
* Subjects with symptoms not consistent with type 1 food reactions (atopic dermatitis, eosinophilic esophagitis and any other non-IgE-mediated food sensitivities) will be excluded.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, beta-blocker use or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Subjects on anticoagulants, anti-platelet therapy, or any other predisposition towards bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Singh, MD, Principal Investigator — Ann & Robert H. Lurie Childrens Hospital; Bruce Bochner, MD, Principal Investigator — Northwestern Feinberg School of Medicine
Locations (1):
- Ann & Robert H. Lurie Childrens Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dispenza MC, Pongracic JA, Singh AM, Bochner BS. Short-term ibrutinib therapy suppresses skin test responses and eliminates IgE-mediated basophil activation in adults with peanut or tree nut allergy. J Allergy Clin Immunol. 2018 May;141(5):1914-1916.e7. doi: 10.1016/j.jaci.2017.12.987. Epub 2018 Jan 31. No abstract available. PMID 29360526

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were excluded if baseline skin prick tests to peanut/tree nuts were all negative.
Groups:
- Ibrutinib: All participants received 420 mg of ibrutinib orally for 2 to 7 days after undergoing baseline screening criteria.
Period: Overall Study
Arm/Group | Ibrutinib
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adults with a confirmed history of IgE-mediated food allergy were enrolled.
Groups:
- All Participants: All participants received ibrutinib after undergoing baseline screening criteria.
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
Skin prick test to peanut and/or tree nuts [Count of Participants; unit: Participants] — Skin prick tests (SPT) to clinically relevant foods were performed at baseline. All SPTs were performed on the volar aspect of the forearm using Quintip devices and commercially purchased extracts and histamine and saline controls. SPTs were measured 15 minutes after prick, and the area was calculated using the largest diameter of wheal and flare. SPTs were considered positive if the wheal was ≥3 mm in diameter. Subjects whose SPTs were all negative were excluded. Subjects with at least one positive SPT were enrolled. Only positive SPTs at baseline were repeated with subsequent visits.
  Participants | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Doses of Ibrutinib for Maximal Suppression of Skin Prick Test Size to Foods
Description: The primary outcome was the number of ibrutinib doses (2, 4, or 7 doses) required to maximally suppress food skin prick reactivity to foods. All participants received 420 mg ibrutinib orally once daily for 2, 4, or 7 doses after undergoing baseline screening criteria. Skin testing to peant and tree nuts was done at baseline and repeated at each visit on days 2, 4, and 7 (corresponding to 2, 4, or 7 doses of ibrutinib).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: doses
Groups:
- Ibrutinib: All participants received 420 mg ibrutinib orally once daily for 2, 4, or 7 doses after undergoing baseline screening criteria.
Arm/Group | Ibrutinib
Number analyzed (Participants) | 6
doses | 2 (0)
Statistical Analysis 1: Comparison: Ibrutinib; Test type: Superiority — Values for grouped data were reported as mean ± SD and were calculated using Graphpad Prism 7 software (La Jolla, CA), which was also used for generating figures and for statistical analyses. Changes in skin test area (wheal and flare) were analyzed at each time point (after 2 doses, 4 doses, etc) using Friedman tests for grouped analysis and Wilcoxon signed rank tests between pairs; p < 0.0001, Wilcoxon (Mann-Whitney) — The above p value reflects the statistical analysis of skin test area between baseline and 2 doses of ibrutinib; Changes in skin test area at each time point were analyzed using Friedman tests for grouped analysis and Wilcoxon signed rank tests between pairs

2. Secondary Outcome: Number of Doses of Ibrutinib for Maximal Suppression of Basophil Reactivity
Description: The primary outcome was to determine the fewest ibrutinib doses (2, 4, or 7 doses) required to suppress basophil reactivity (BAT). All participants received 420 mg ibrutinib orally once daily for 2, 4, or 7 doses after undergoing baseline screening criteria. Basophil activation testing was perfmored at baseline and repeated at each visit on days 2, 4, and 7 (corresponding to 2, 4, or 7 doses of ibrutinib).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Ibrutinib
Number analyzed (Participants) | 6
doses | 2 (0)
Statistical Analysis 1: Comparison: Ibrutinib; Test type: Superiority — Changes in BAT were analyzed at each time point (after 2 doses, 4 doses, etc) using repeated measures ANOVA for grouped analysis and paired Students t tests between pairs. A p value < 0.05 was considered significant; p < 0.001, ANOVA — The above p value reflects the statistical analysis of BAT between baseline and 2 doses of ibrutinib; Changes in BAT were analyzed at each time point using repeated measures ANOVA for grouped analysis and paired Students t tests between pairs

3. Secondary Outcome: Time to Recovery of Skin Test Reactivity
Description: Another secondary outcome was to determine the timing of when skin prick testing (SPT) response to peanut or tree nuts returned to baseline compared to basophil activation test (BAT) responses. Participants underwent SPT and BAT weekly after cessation of ibrutinib therapy. SPT and BAT that were ≥80% of baseline values were considered to have "returned to baseline."
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- Ibrutininb: All participants received 420 mg ibrutinib orally once daily for 2, 4, or 7 days after undergoing baseline screening criteria.
Arm/Group | Ibrutininb
Number analyzed (Participants) | 6
weeks | 1.24 (0.6633)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over a period of 4 months for each participant - this covers the time from enrollment (and baseline screening procedures) to the 3 month follow-up visit which included laboratory testing for potential toxicity.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=6)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (6) — 1 participant complained of shortness of breath and throat tightness 4 hours after skin prick testing to foods was performed at a scheduled follow-up visit (7 days after completion of the study drug).
Nausea (Gastrointestinal disorders) | 1 (6) — 1 participant had transient nausea with ibrutinib doses 1 and 3, but not with any other doses out of a total 7-day course.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT03149315/Prot_SAP_001.pdf
  • Informed Consent Form (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT03149315/ICF_000.pdf